CLINICAL TRIAL: NCT05509075
Title: Valutazione Dell'Efficacia e Della Sicurezza Dei Nutraceutici Utilizzati Nella Popolazione Generale Per il Trattamento di Patologie Sistemiche o Locali
Brief Title: Nutraceuticals and Functional Foods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Sanitaria Provinciale Di Catanzaro (Other); Azienda Ospedaliera Universitaria Policlinico (Other); Azienda Ospedaliera Pugliese Ciaccio (Other); Annunziata Hospital, Cosenza, Italy (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Prof, University of Catanzaro
Other Study IDs: Nutraceuticals
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Systemic Disease; Skin Diseases; Memory Disorders; Urologic Diseases; Gastrointestinal Diseases; Inflammatory Disease; Pain, Acute; Pain, Chronic; Infective Disorder; Immune System Diseases; Immune Defect
Keywords: systemic diseases; topic diseases; nutrients
MeSH Terms: conditions — Skin Diseases; Memory Disorders; Urologic Diseases; Gastrointestinal Diseases; Acute Pain; Chronic Pain; Communicable Diseases; Immune System Diseases | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- nutraceuticals and neurological disorders: evaluation of nutraceuticals in subjects with memory disorders
  Interventions: Dietary Supplement: nutraceuticals
- nutraceuticals and skin disorders: evaluation of nutraceuticals in clinical conditions requiring topical treatment for skin diseases
  Interventions: Dietary Supplement: nutraceuticals
- nutraceuticals and gastrointestinal diseases: evaluation of nutraceuticals in clinical conditions requiring systemic treatment for gastrointestinal diseases
  Interventions: Dietary Supplement: nutraceuticals
- nutraceuticals and urological diseases: evaluation of nutraceuticals in the management of patients with prostate diseases or with lower tract infectious diseases requiring systemic or local treatment
  Interventions: Dietary Supplement: nutraceuticals
- nutraceuticals and immunomediate diseases: evaluation of nutraceuticals in the management of patients with immunomediate disorders
  Interventions: Dietary Supplement: nutraceuticals
- nutraceuticals and pain: evaluation of nutraceuticals in the management of patients with acute or chronic pain
  Interventions: Dietary Supplement: nutraceuticals

INTERVENTIONS:
Dietary Supplement: nutraceuticals — antioxidants

SUMMARY:
Supplements and functional foods are now readily available and usable by the general population. Many supplemnets are commonly used in poly-treated patients where interactions or adverse events may develop, therefore we evaluate in the rela life the use of nutraceuticals, their clinical effects and the development of adverse drug reactions

DETAILED DESCRIPTION:
Supplements (also called nutraceuticals because they derive from natural substances) and functional foods are now readily available and usable by the general population. The term "nutraceutical" derives from a fusion of the terms "nutritional" and "pharmaceutical" y was used for the first time in 1989 by Stephen De Felice, President of the Fundación para la Innovación en Medicine (Cranford, NJ, EE. UU. ). On the other hand, functional foods have additional effects due to the presence of components, generally non-nutritious, which interact selectively with one or more physiological functions of the organism (biomodulation) in such a way that an improvement in the state of health and well-being is evident. And/or a reduced risk of disease.

The Regulation EC / 178/2002 of the Parliament and the Council, 28/01/2002 establishes the general principles and requirements of food law, shows the European Food Safety Authority (EFSA), and establishes the procedures in the field of food safety.

Given their documented efficacy following the European Claims, which indicate for each substance what the individual uses may be (EFSA Journal 2011; 9 (4): 1984; EFSA Journal 2011; 9 (4): 2061; EFSA Journal 2012 ; 10 (3): 2604; EFSA Journal 2012; 10 (5): 2702; EFSA Journal 2016; 14 (1): 4367; EFSA Journal 2017; 15 (1): 4680; EFSA Journal 2018; 16 (1): 5136), a doubt related to safety in the general population remains today.

For this reason, in the month of March 2018, the Health and Quality of Life Working Group of the Italian Federation of Life Sciences (Fisv), which also includes the Italian Society of Pharmacology (Sif), the Italian Anthropological Association (Aai), Italian Agricultural Chemistry (Sica), Italian Society of Environmental Mutagenesis (Sima), Italian Society of General Microbiology and Microbial Biotechnology (Simgbm) and Italian Society of Plant Pathology (Sipav) has re-evaluated the scientific bibliography on the use of supplements or supplements food and has assessed that in the vast majority of cases their use is not only improper - as a good diet would be much more efficient to "heal" any deficiencies in trace elements or vitamins - but that often these products can cause undesirable effects, both for the concomitance of pathologies or pharmacological treatments with which they can interfere, both for the potential toxicity and oligopoly Minds and vitamins can exert on the body if their level of intake is higher than the needs of the moment. This is because many if not all of these supplements are authorized without having objective clinical safety data. Many of these are also used in poly-treated patients where interactions or adverse events may develop that are underestimated or unrecognized.

In consideration of the fact that the nutraceutical market is constantly growing (it is estimated 90 thousand products for over 30 billion dollars in turnover only in the US and 3 in Italy.), The need arises to evaluate "real life" in a manner objective to the possible efficacy and safety of nutraceuticals and functional foods used to treat systemic or local diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients or healthy subjects of both sexes and aged> 18 years Patients are not on supplement therapy or functional foods for any purpose.
* Patients who have given their consent to participate in the study

Exclusion Criteria:

* Patients with severe renal or liver failure, neoplastic diseases or those with allergy to supplement or functional food , and those who do not sign the consent will be excluded from the study. Informed.

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At admission (T0), the anthropometric data and the functional clinical data of each patient (or healthy subject) will be collected. An aliquot of the blood sample will be used for transcriptomic evaluation.
  Immediately after the clinical and laboratory evaluation, each GP or each specialist will decide the type of nutraceutical or functional food to be used. For example, in elderly patient with osteoarthritis disorders can use a supplement based on chondroitin or glucosamine or other substances (or functional foods) with specific claims, as well as a patient with hypercholesterolemia without other risk factors can use a supplement containing monacolin K or flavonoids or other functional foods with claims specific. Similarly, patients with gastrointestinal or genitourinary disorders can use functional food based on probiotics or substances with a particular activity and comply with international claims.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
improvement of memory | 6 months
  Mini-mental state examination: range from 0 (worst) to 30 (no deficit) (< 18 severe deficit, 19-24 mild deficit, >25 normal function)
improvement of pain | 6 months
  Visual analogical scale: range from 0 (no pain) to 10 (high pain) > 8 severe pain; 4-7 moderate pain; 1-3 mild pain)

SECONDARY OUTCOMES:
change in plasma lipid values | 12 months
  LDL (mg/dL), HDL (mg/dL), total cholesterol (mg/dL)
improvement of quality of life | 6 months
  36-Item Short Form Health Survey (SF-36), range from 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Luca Gallelli, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaccaro MG, Innocenti B, Cione E, Gallelli L, De Sarro G, Bonilla DA, Cannataro R. Acute effects of a chewable beetroot-based supplement on cognitive performance: a double-blind randomized placebo-controlled crossover clinical trial. Eur J Nutr. 2024 Feb;63(1):303-321. doi: 10.1007/s00394-023-03265-y. Epub 2023 Oct 24. PMID 37875637